CLINICAL TRIAL: NCT02360943
Title: Pharmacoepidemiology Treatment of Symptomatic Pulmonary Embolism in Hospitalized Patients Aged 75 Years or More: Prospective, Multicenter Cohort Study PEAGE
Brief Title: Pharmacoepidemiology Treatment of Symptomatic Pulmonary Embolism in Hospitalized Patients Aged 75 Years or More: PEAGE
Acronym: PEAGE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 1208182; 2013-000315-24 (EudraCT Number)
Record Dates: First submitted 2015-02-06; First posted 2015-02-11 (Estimated); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Elderly; Pulmonary Embolism; Anticoagulants
Keywords: elderly patients; Pulmonary embolism; Anticoagulant treatments
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PEAGE: Patients older than 75 years receiving an anticoagulant treatment for a symptomatic and confirmed PE
  Interventions: Other: 4 blood samples

INTERVENTIONS:
Other: 4 blood samples — PK and / or PD measurements during hospitalization

SUMMARY:
The treatment of the venous thromboembolic disease, including pulmonary embolism (PE), is based on anticoagulants. During the last decade, all the randomized clinical trials evaluating these anticoagulants have included PE patients with an average age below 60 years. But in clinical pratice, approximately 50% of PE patients are older than 75 years.

So the investigators want to perform a french multicentre prospective cohort of consecutive patients receiving an anticoagulant treatment for a symptomatic and confirmed PE. All the validated and available anticoagulant treatments are authorized in this cohort (unfractionnated and low molecular weight heparins, fondaparinux, vitamin K antagonists and direct oral anticoagulants).

This cohort will provide data regarding the bleeding risk and the risk of PE recurrences and regarding the pharmacokinetic (PK) and pharmacodynamic (PD) properties of these anticoagulants in this older population. Using population approach modelling , the investigators will pay particular attention to the sources of PK/PD variability PK / PD such as genetic polymorphisms of P-glycoprotein and cytochrome P450.

Using all these data , the investigators will try to identify significant risk factors for bleeding and venous thromboembolic events.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic pulmonary embolism confirmed by objective paraclinical examination with or without DVT associated
* confirmation of pulmonary embolism within 3 days
* Administration possible according to the recommended dosages of anticoagulant treatment : (unfractionnated and low molecular weight heparins, fondaparinux, vitamin K antagonists and direct oral anticoagulants)
* Indication of anticoagulant treatment for at least 6 months

Exclusion Criteria:

* on therapeutic dose of anticoagulant treatment over 72 hours
* indication to therapeutic dose of anticoagulant treatment for another reason.
* Inability for whatever reasons, to prescribe recommended anticoagulant treatment
* PE treatment on heparin-induced thrombocytopenia requiring argatroban, lepirudin or danaparoid treatment,
* ongoing bleeding
* PE occurring despite well conducted anticoagulant treatment
* Contraindications to recommended dose of anticoagulant treatment

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: patients older than 75 years receiving an anticoagulant treatment (unfractionnated and low molecular weight heparins, fondaparinux, vitamin K antagonists and direct oral anticoagulants) for a symptomatic and confirmed pulmonary embolism
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2014-07-09 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2022-04-22 (Actual)

PRIMARY OUTCOMES:
Major bleeding defined by the International Society of Thrombosis & Haemostasis | at 6 months
  * Bleeding causing a fall in hemoglobin level of 20 g L-1 (1.24 mmol L-1) or more, or leading to transfusion of two or more units of whole blood or red cells.,
  * Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intra-articular or pericardial, or intramuscular with compartment syndrome,
  * Fatal bleeding

SECONDARY OUTCOMES:
Clinically relevant non-major bleeding | at 6 months
  defined by:
  * Subcutaneous hematoma spontaneous over 25 cm2
  * Spontaneous epistaxis for more than 5 minutes
  * Spontaneous or after urinary catheter hematuria for more than 24 hours
  * Significant rectal bleeding
  * Gingival bleeding for more than 5 minutes
  * Bleeding requiring hospitalization and / or a hemostatic action
Recurrent pulmonary embolism | at 6 months
  confirmed by CT scan or ventilation/perfusion lung scan
Deep vein thrombosis (recurrence or new) | at 6 months
  confirmed by venous doppler ultrasonography or venography of the lower limbs or CT scan
Arterial cardiovascular events | at 6 months
  * Acute coronary syndrom with or without ST-segment elevation
  * Stroke ischemic or hemorrhagic confirmed by CT scan or magnetic resonance imaging brain
  * Acute ischemic phenomena (lower limbs, mesenteric ...) confirmed by arterial doppler or arteriography.
Death | at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Patrick MISMETTI, MD PhD, Principal Investigator — CHU de Saint Etienne
Locations (20):
- France (20):
  - CHU d'Angers, Angers
  - Hôpital Universitaire Jean Minjoz, Besançon
  - CHU de Brest, Brest
  - Clinique du Parc - Castelnau Le Lez, Castelnau-le-Lez
  - CHU Gabriel Montpied, Clermont-Ferrand
  - Hôpitaux Universitaires Louis Mourier Paris Nord, Colombes
  - CHU de Dijon, Dijon
  - CHU de Grenoble, Grenoble
  - CHU de Limoges, Limoges
  - CHU de Montpellier, Montpellier
  - CHRU de Nantes, Nantes
  - CHU de Nice, Nice
  - Hôpital Europeen Georges Pompidou, APHP, Paris
  - APHP Hôpital BROCA, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU de Rouen, Rouen
  - CHU de Saint Etienne, Saint-Etienne
  - CHU de Strasbourg - Hôpital Civil, Strasbourg
  - Centre Hospitalier Intercommunal Toulon La Seyne sur Mer, Toulon
  - CHU Tours, Tours

IPD SHARING:
Plan to Share IPD: No